CLINICAL TRIAL: NCT04765280
Title: Evaluation of the Relationship Between Central Sensitization and Disability in Patients With Chronic Musculoskeletal Pain in Physical Medicine and Rehabilitation Clinic.
Brief Title: The Frequency of Central Sensitization in Patients With Chronic Musculoskeletal Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.114
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-11

CONDITIONS: Central Sensitisation; Chronic Musculoskeletal Disease; Chronic Pain
Keywords: central sensitization; central sensitization inventory; disability; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic musculoskeletal pain: Patients with any musculoskeletal pain for at least 3 months
  Interventions: Diagnostic Test: Central sensitization inventory; Other: Short form-36; Other: Istanbul Low Back Pain Disability Index; Other: Disabilities of the Arm, Shoulder and Hand (DASH); Other: Neck Pain and Disability scale; Other: Knee Injury and Osteoarthritis Outcome Score; Other: Western Ontario and McMaster Universities Arthritis Index; Other: Visual analogue scale

INTERVENTIONS:
Diagnostic Test: Central sensitization inventory — Standardized questionnaire to determine the level of central sensitization. Patients with a score of 40 and above are considered to have central sensitization.
  Other Names: CSI
Other: Short form-36 — Standardized questionnaire to investigate the quality of life in patients. The score of the scale is between 0-100. The higher scores are associated with greater deterioration in quality of life.
  Other Names: SF-36
Other: Istanbul Low Back Pain Disability Index — Standardized questionnaire to investigate the disability in patients with low back pain. The score of the scale is between 0-90. It is accepted that the higher the score, the higher the disability.
  Other Names: ILBPDI
Other: Disabilities of the Arm, Shoulder and Hand (DASH) — Standardized questionnaire to investigate the disability in patients with upper extremity musculoskeletal disorders. The score of the scale is between 0-100 It is accepted that the higher the score, the higher the disability.
  Other Names: Quick DASH
Other: Neck Pain and Disability scale — Standardized questionnaire to investigate the disability in patients with neck pain. The score of the scale is between 0-100. It is accepted that the higher the score, the higher the disability.
  Other Names: NPAD
Other: Knee Injury and Osteoarthritis Outcome Score — Standardized questionnaire to investigate the disability in patients with knee pain. The score of the scale is between 0-100It is accepted that the higher the score, the higher the disability.
  Other Names: KOOS
Other: Western Ontario and McMaster Universities Arthritis Index — Standardized questionnaire to investigate the disability in patients with hip osteoarthritis. The score of the scale is between 0-240. It is accepted that the higher the score, the higher the disability.
  Other Names: WOMAC
Other: Visual analogue scale — global pain score on a 0 to 10
  Other Names: VAS

SUMMARY:
Central sensitization is as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with in many musculoskeletal diseases with chronic pain has been demonstrated in several studies. However, the effect of central sensitization on disability in these patients is not fully known. In this study, it was aimed to investigate the frequency of central sensitization and its effect on patients with chronic musculoskeletal pain who were admitted to physical medicine and rehabilitation outpatient clinics.

DETAILED DESCRIPTION:
The term central sensitization (CS) was first used in 1988 and was explained as the increase in pain sensitivity with the amplification of neuron-derived signals in the central nervous system. With the development of CS, a decrease in the pain threshold and an increase in generalized sensitivity occur. There is no method for the diagnosis of CS is accepted as a gold standard. Clinical scales and quantitative sensory testing (QST) is used for this purpose widely. In addition, the well-known scale used for the evaluation of CS is the Central Sensitization Inventory (CSI), developed for detect CS in chronic pain patients. The use of CSI, which is more practical to use, is becoming widespread because QST takes time, is costly and requires experienced practitioners. The prevalence of chronic pain is reported as 30% in Europe and has an important place among diseases that cause disability worldwide. Until this time, the relationship between CS and many diseases that cause chronic pain has been revealed, and an increase in pain intensity, duration and prevalence has been detected in patients accompanied by CS. In addition to all these changes, the decrease in the treatment response of these patients makes the clinical management of individuals with pain sensitization even more difficult. Although the increase in the frequency of CS in patients with chronic pain is known, data on the incidence of this condition in various diseases with chronic pain is limited.The frequency of CS was mostly reported in patients with low back (37.8%) and neck pain (32.4%) and the authors reported that the higher rates of disability is seen in patients with high CSI scores. Similarly, in this study, it was planned to show the relationship between CS and disability in patients with chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Have musculoskeletal pain that lasts for at least 3 months
* Accepting to participate in the study

Exclusion Criteria:

* Have rheumatic disease

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients aged 18-75 years diagnosed with chronic musculoskeletal disorders will be recruited from a PMR outpatient clinic of a state hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | 6 months
  25 somatic and psychosocial symptoms, which are frequently found in patients with central sensitization in part A, are questioned. In part B, the presence of diseases whose relationship with central sensitization is well defined is questioned in the patient without participating in scoring. Central sensitization is assumed in patients who score 40 or more over 100 points.

SECONDARY OUTCOMES:
VAS pain | 6 months
  The patients pain severity will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
SF-36 | 6 months
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health.The scale was developed by Ware in 1987 and consists of 36 questions questioning 8 sub-parameters regarding the health status of the person.These parameters are physical function, pain, limitation due to physical and emotional problems, emotional well-being, social function, fatigue and general health perception.
Istanbul Low Back Pain Disability Index (ILBPDI) | 6 months
  This scale was developed for assessing the severity of disability in chronic low back pain patients by Duruöz et.al in 2013. This scale consists of 18 questions in the form of a Likert scale that evaluates the limitation of daily life activities of patients in the last month.It is accepted that the higher the score, the higher disability.
The Neck Pain and Disability scale (NPAD) | 6 months
  The NPAD is a composite index including 20 items which measure the intensity of neck pain and related disability.It is accepted that the higher the score, the higher disability
Quick DASH | 6 months
  The Quick DASH is a shortened version of the questionnaire, which was created to detect symptoms and loss of function secondary to musculoskeletal problems of the upper extremity.There are 30 questions in the original form of the questionnaire, and the newly developed short version has been reduced to 11 questions in total. Beaton et al stated that with the quick questionnaire for arm, shoulder and hand problems, upper extremity functional evaluation can be made at rates similar to the original version.
KOOS | 6 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
WOMAC | 6 months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain, stiffness and physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Canan ŞANAL TOPRAK, Asst.Prof, Study Chair — Marmara University
Locations (1):
- Feyza Nur YUCEL, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Woolf CJ, Thompson SW, King AE. Prolonged primary afferent induced alterations in dorsal horn neurones, an intracellular analysis in vivo and in vitro. J Physiol (Paris). 1988-1989;83(3):255-66. PMID 3272296
- [Result] Gervais-Hupe J, Pollice J, Sadi J, Carlesso LC. Validity of the central sensitization inventory with measures of sensitization in people with knee osteoarthritis. Clin Rheumatol. 2018 Nov;37(11):3125-3132. doi: 10.1007/s10067-018-4279-8. Epub 2018 Sep 3. PMID 30178171
- [Result] Nijs J, Malfliet A, Ickmans K, Baert I, Meeus M. Treatment of central sensitization in patients with 'unexplained' chronic pain: an update. Expert Opin Pharmacother. 2014 Aug;15(12):1671-83. doi: 10.1517/14656566.2014.925446. Epub 2014 Jun 15. PMID 24930805
- [Result] Roldan-Jimenez C, Perez-Cruzado D, Neblett R, Gatchel R, Cuesta-Vargas A. Central Sensitization in Chronic Musculoskeletal Pain Disorders in Different Populations: A Cross-Sectional Study. Pain Med. 2020 Nov 1;21(11):2958-2963. doi: 10.1093/pm/pnaa069. PMID 32232473
- [Result] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Result] Tanaka K, Murata S, Nishigami T, Mibu A, Manfuku M, Shinohara Y, Tanabe A, Ono R. The central sensitization inventory predict pain-related disability for musculoskeletal disorders in the primary care setting. Eur J Pain. 2019 Oct;23(9):1640-1648. doi: 10.1002/ejp.1443. Epub 2019 Aug 1. PMID 31233655
- See also: Neck pain and disability scale — https://www.physio-pedia.com/Neck_Pain_and_Disability_Scale
- See also: SF-36 — https://www.physio-pedia.com/36-Item_Short_Form_Survey_(SF-36)
- See also: KOOS — https://www.physio-pedia.com/Knee_Injury_and_Osteoarthritis_Outcome_Score